CLINICAL TRIAL: NCT05308537
Title: The Effectiveness of the Mindful Compassion Care Program (MCCP) in Reducing Burnout and Psychological Distress Amongst Frontline Hospital Nurses During the COVID-19 Pandemic: a Randomized Controlled Trial
Brief Title: Randomized Controlled Trial of the Mindful Compassion Care Program in Reducing Psychological Distress Amongst Nurses During the COVID-19 Pandemic
Acronym: MCCP-COVID19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Antonio Lasalvia, Principal Investigator, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3717CESC
Record Dates: First submitted 2022-04-01; First posted 2022-04-04 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Burnout; COVID-19
Keywords: mindfulness; compassion; burnout; emotional exhaustion; COVID-19; healthcare workers; nurse
MeSH Terms: conditions — Burnout, Psychological; COVID-19; Emotional Exhaustion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Compassion Care Program (Experimental): The MCCP comprises six regular 1 hour and 30-minute sessions and 1 all-day class lasting 4 hours and 30 minutes.
  Interventions: Behavioral: Mindful Compassion Care Program
- Waiting List (No Intervention)

INTERVENTIONS:
Behavioral: Mindful Compassion Care Program — The intervention is a proven effective mindfulness programme based on well-known scientific programmes such as mindfulness-based stress reduction mindfulness-based cognitive therapy and compassion focused therapy.
  Arms: Mindful Compassion Care Program

SUMMARY:
Recent studies have shown that nurses have been more affected by the COVID-19 pandemic than any other group of hospital workers in terms of anxiety, depression, and burnout. Several clinical studies had previously demonstrated the effectiveness of mindfulness and compassion interventions in reducing burnout and emotional distress amongst healthcare professionals. A parallel-group randomized controlled trial will assess the feasibility, acceptability, and efficacy of a mindfulness and compassion-focused programme on frontline nurses who had been working during the COVID-19 pandemic. Seventy-two participants will be divided equally into an intervention group and a control group. Primary outcome will be assessed using the Emotional Exhaustion subscale of the Maslach Burnout Inventory General Survey (MBI-GS). Secondary outcomes will be measured by the Cynicism and Professional Efficacy subscales of the MBI-GS; the Patient Health Questionnaire (PHQ-9); the Generalized Anxiety Disorder (GAD-7); the Insomnia Severity Index (ISI); the Impact of Stressful Events (IES-R); the Perceived Stress Scale (PSS); the Five Facet Mindfulness Questionnaire (FFMQ); and the Forms of Self-Criticising/attacking and Self-Reassuring Scale (FSCRS). The study aims to fill a gap in the literature and present a scientifically validated intervention for those healthcare professionals most exposed to the stressful conditions of working during the COVID-19 pandemic.

DETAILED DESCRIPTION:
BACKGROUND. From the beginning of the COVID-19 pandemic, healthcare workers (HCWs) worldwide experienced overwork, increased health risks in the absence of clear guidelines, and the reorganisation of their activities. These factors, combined with exposure to a condition of increased mortality and a sense of uncontrollability, have led to growing incidences of burnout, anxiety, depressive symptoms, and a reduced investment of energy in the professional sphere. Nurses were amongst the HCWs most exposed to the negative psychological effects of the COVID-19 pandemic, particularly those working in departments most involved in the treatment of COVID-19 patients, such as intensive care, infectious disease, and pulmonary units and emergency rooms. Several studies have shown the effects of mindfulness interventions in reducing burnout and emotional distress among HCWs in the pre-COVID 19 era. Mindfulness can be defined as an awareness of present-moment thoughts, feelings, and bodily sensations through intentional and non-judgemental attention. It is a state of consciousness that allows the mind and body to build a relationship of harmony and balance, a predisposing element for the condition of well-being. Studies investigating the diffusion of clinical models based on mindfulness have allowed us to hypothesize that it can play an important role in emotional self-regulation. It can, therefore, be argued that mindfulness allows one to reduce suffering and create a healthy mind by using self-processing processes and modulating awareness of self and one's emotional states, behaviours, as well as relationships with others. The ability to manage suffering, for example of patients and caregivers, stems from an empathic and emotional attunement known as compassion to the suffering of the another person. Compassion can be defined as the awareness of one's own and others' suffering and the intention or motivation to alleviate it. It has been associated with the capacity to adjust to distressful experiences during dramatic events such as pandemics, and amongst HCWs in particular.

AIMS. Studies evaluating the efficacy of mindfulness among HCWs s working during the current COVID-19 pandemic are rare, though some are in progress. The present project is based on the results of a longitudinal study that assessed the psychological impact of the COVID-19 pandemic on HCWs at the Verona University Hospital Trust during the lockdown phase and after one year later. The present project proposed here aims to implement and evaluate the feasibility, acceptability, and effectiveness of a preliminarily tested intervention that integrates the most widely used and scientifically validated mindfulness protocols such as mindfulness-based stress reduction, mindfulness-based cognitive therapy, and compassion focused therapy, in a healthcare context (the Verona University Hospital Trust) during the COVID-19 pandemic. The purpose of the intervention is to reduce burnout and psychological distress among frontline nurses involved in the clinical management of COVID-19 patients. The study will be conducted at the Verona University Hospital Trust (Azienda Ospedaliera Universitaria Integrata [AOUI]), the second-largest hospital in Italy in terms of the number of beds and the fifth largest in terms of admissions. The trust employs 6,000 people, including nearly 2,000 nurses. On 17 March 2020, the Veneto regional government converted part of the hospital into a COVID-19 hospital. Dedicated pathways for both suspected and confirmed COVID-19 cases were established within the hospital, as well as in other hospital units located in clearly restricted areas devoted to the treatment of COVID-19 patients.

DESIGN. Participants will be randomly assigned to one of two groups: the experimental group will receive the Mindful Compassion Care Program (MCCP), and the control group will be allocated to a waiting list (WL). The effectiveness of the experimental intervention will be assessed by comparing the changes in the level of burnout at the end of the treatment and after 1-month later. Other psychological dimensions will also be investigated (i.e., anxiety and depressive symptoms, post-traumatic symptoms, insomnia, perception of stress, mindfulness skills and evaluation of self-criticism and self-reassurance).

Enrollment procedure: The study description and the invitation to participate will be published in the hospital's newsletter and will be emailed to the nurses' address by the Verona Hospital Trust Administration. All nurses who express an interest in participating will receive (via email) an information sheet containing all the project details together with a link to the online screening questionnaire. They will find the participant consent form and the consent form for the use and processing of personal data on the same page. The screening questionnaire will allow us to assess whether the participant meets the inclusion criteria. If they do, they will be added to a temporary list of candidates; if they do not, they will be excluded from the trial. Participants will be randomly allocated to the intervention or the WL control group with an allocation ratio of 1:1. Participants allocated to the experimental group will receive the intervention immediately after randomization, and those assigned to the control group will be offered the same intervention 6 months after. The experimental intervention will take place over 6-weeks. The pre-test, post-test, and 1-month follow-up will be carried out at the same time for both study groups. The trial will begin in April 2022. Enrolment will end as soon as the expected number is reached (36 for the intervention group and 36 for the control group). Before the intervention, participants randomly assigned to the intervention group will be divided into three subgroups consisting of 12 individuals. Each subgroup will follow the mindfulness courses (led by the same instructor) for 6 weeks. The courses will be delivered every Monday for subgroup 1, Tuesday for subgroup 2, and Wednesday for subgroup 3. Nurses will attend the intervention during working hours as part of the continuing professional education (CPE) courses provided by the Verona Hospital Trust Administration.

BASELINE ASSESSMENT. Before entering the study, participants screening positive will be asked to provide informed consent to participate. Primary outcome will be assessed using the Emotional Exhaustion subscale of the Maslach Burnout Inventory General Survey (MBI-GS). Secondary outcomes will be measured by the Cynicism and Professional Efficacy subscales of the MBI-GS; the Patient Health Questionnaire (PHQ-9); the Generalized Anxiety Disorder (GAD-7); the Insomnia Severity Index (ISI); the Impact of Stressful Events (IES-R); the Perceived Stress Scale (PSS); the Five Facet Mindfulness Questionnaire (FFMQ); and the Forms of Self-Criticising/attacking and Self-Reassuring Scale (FSCRS).

FOLLOW-UP ASSESSMENT. After 1 months from the end of the intervention participants will be re-assessed for Emotional Exhaustion subscale of the Maslach Burnout Inventory General Survey (MBI-GS). Secondary outcomes will be measured by the Cynicism and Professional Efficacy subscales of the MBI-GS; the Patient Health Questionnaire (PHQ-9); the Generalized Anxiety Disorder (GAD-7); the Insomnia Severity Index (ISI); the Impact of Stressful Events (IES-R); the Perceived Stress Scale (PSS); the Five Facet Mindfulness Questionnaire (FFMQ); and the Forms of Self-Criticising/attacking and Self-Reassuring Scale (FSCRS).

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, a participants will have to be:

* a nurse employed at AOUI for the past two years;
* working within intensive care units, infectious disease unit, pulmonary medicine and internal medicine units that have been converted to COVID-19 sub-intensive units;
* scoring above the cut-off score for the Emotional Exhaustion sub-scale (EX) of the MBI-GS (equal to or greater than 2.20) in accordance with Italian norms

Exclusion Criteria:

Respondents will be excluded if they:

* have participated in mindfulness-based interventions in the previous 6 months;
* show a score < 2.20 in the EX subscale of the MBI-GS;
* are receiving psychosocial or psychiatric treatment. Participants allocated to the WL will be requested not to participate in a mindfulness course offered elsewhere.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-02-19 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Emotional exhaustion | Change from baseline at 1 month follow-up
  Emotional exhaustion (EX) is a psychological construct that explores the perception of physical and emotional fatigue. It is characterized specifically by a lack of energy required to handle daily life and the prevalence of feelings of apathy and emotional detachment at work. EX is measured through the use of the Maslach Burnout Inventory-General Survey. The items were scored on a Likert scale from 0 (never) to 6 (everyday) (Schaufeli et al. 1996). High score is indicative of high levels of burnout.

SECONDARY OUTCOMES:
Personal socio-demographic information | Baseline
  These information will be collected by using an ad hoc schedule, addressing personal and job-related characteristics.
Professional efficacy and cynicism | Change from baseline at 1 month follow-up
  Maslach Burnout Inventory-General Survey. Cynicism (5 items), which measures an indifference or a distant attitude towards your work; professional efficacy (6 items), which measures satisfaction with past and present accomplishments, and it explicitly assesses an individual's expectations of continued effectiveness at work. The items were scored on a Likert scale from 0 (never) to 6 (everyday) (Schaufeli et al. 1996). High score is indicative of high levels of burnout.
Depressive symptoms | Change from baseline at 1 month follow-up
  Patient Health Questionnaire (PHQ-9) that is a nine-question self-report measure. Respondents are asked how much each symptom has bothered them over the past 2 weeks, with response options of "not at all", "several days", "more than half the days", and "nearly every day", scored as 0, 1, 2, and 3. The scale can range from 0 to 48, with higher scores indicating higher levels of depression and anxiety symptomatology.
Anxiety symptoms | Change from baseline at 1 month follow-up
  Generalized Anxiety Disorder (GAD-7) is a self-rated questionnaire consisting of seven items that investigate the level of anxiety and worry. The GAD-7 scale score ranges from 0 to 21 points. A score between 5 and 9 points characterizes mild GAD. Between 10 and 14, moderate GAD and between 15 and 21, severe GAD.
Insomnia | Change from baseline at 1 month follow-up
  Insomnia Severity Index (ISI) is a seven-item questionnaire that asks respondents to rate the nature and symptoms of their sleep problems. Each item is scored 0 (no problem) - 4 (very big problem) with total between 0-28 (absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Post-traumatic symptoms | Change from baseline at 1 month follow-up
  Impact of Events Scale - Revised version (IES-R) is a 22-item self-report that assesses subjective distress caused by traumatic events. Range 0-88. Higher scores mean worse outcome.
Perception of stress | Change from baseline at 1 month follow-up
  Perceived Stress Scale (PSS) is a 10-item questionnaire to measure the degree to which life situations are appraised as stressful. It is a 10-item scale, with a total range from 0 (no symptoms) to 40 (highest severity).
Mindfulness skills | Change from baseline at 1 month follow-up
  The Five Facet Mindfulness Questionnaire (FFMQ) is a self-report measure consisting of 39 items based on a five-facet model (i.e., observe, describe, act with awareness, nonjudgement, and nonreaction) The possible score ranged from 1-5. Higher scores indicate a greater level of mindfulness.
Evaluation of self-criticism and self-reassurance | Change from baseline at 1 month follow-up
  Forms of Self-Criticising/attacking and Self-Reassuring Scale (FSCRS) is a self-administered tool for the assessment of three forms of self-to-self relating as a process measure. The FSCRS is a 22-item self-report questionnaire in which participants are asked to rate how they typically think and react when things go wrong for them. To a first probe statement, 'When things go wrong for me…', participants responded on a 5-point Likert scale (ranging from 0 = not at all like me to 4 = extremely like me). Higher scores indicate a higher level of self-criticism.

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Verona, Verona, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lasalvia A, Amaddeo F, Porru S, Carta A, Tardivo S, Bovo C, Ruggeri M, Bonetto C. Levels of burn-out among healthcare workers during the COVID-19 pandemic and their associated factors: a cross-sectional study in a tertiary hospital of a highly burdened area of north-east Italy. BMJ Open. 2021 Jan 17;11(1):e045127. doi: 10.1136/bmjopen-2020-045127. PMID 33455940
- [Background] Lasalvia A, Bonetto C, Porru S, Carta A, Tardivo S, Bovo C, Ruggeri M, Amaddeo F. Psychological impact of COVID-19 pandemic on healthcare workers in a highly burdened area of north-east Italy. Epidemiol Psychiatr Sci. 2020 Dec 17;30:e1. doi: 10.1017/S2045796020001158. PMID 33331255
- [Background] Lasalvia A, Bodini L, Amaddeo F, Porru S, Carta A, Poli R, Bonetto C. The Sustained Psychological Impact of the COVID-19 Pandemic on Health Care Workers One Year after the Outbreak-A Repeated Cross-Sectional Survey in a Tertiary Hospital of North-East Italy. Int J Environ Res Public Health. 2021 Dec 19;18(24):13374. doi: 10.3390/ijerph182413374. PMID 34948981
- [Background] La Torre G, Raffone A, Peruzzo M, Calabrese L, Cocchiara RA, D'Egidio V, Leggieri PF, Dorelli B, Zaffina S, Mannocci A, Yomin Collaborative Group. Yoga and Mindfulness as a Tool for Influencing Affectivity, Anxiety, Mental Health, and Stress among Healthcare Workers: Results of a Single-Arm Clinical Trial. J Clin Med. 2020 Apr 7;9(4):1037. doi: 10.3390/jcm9041037. PMID 32272758
- [Background] Matos M, McEwan K, Kanovsky M, Halamova J, Steindl SR, Ferreira N, Linharelhos M, Rijo D, Asano K, Marquez MG, Gregorio S, Vilas SP, Brito-Pons G, Lucena-Santos P, da Silva Oliveira M, de Souza EL, Llobenes L, Gumiy N, Costa MI, Habib N, Hakem R, Khrad H, Alzahrani A, Cheli S, Petrocchi N, Tholouli E, Issari P, Simos G, Lunding-Gregersen V, Elklit A, Kolts R, Kelly AC, Bortolon C, Delamillieure P, Paucsik M, Wahl JE, Zieba M, Zatorski M, Komendzinski T, Zhang S, Basran J, Kagialis A, Kirby J, Gilbert P. Compassion Protects Mental Health and Social Safeness During the COVID-19 Pandemic Across 21 Countries. Mindfulness (N Y). 2022;13(4):863-880. doi: 10.1007/s12671-021-01822-2. Epub 2022 Jan 4. PMID 35003380
- [Background] Cheli S, De Bartolo P, Agostini A. Integrating mindfulness into nursing education: A pilot nonrandomized controlled trial. Int J Stress Manag. 2020;27(1):93.
- [Derived] Bodini L, Bonetto C, Cheli S, Del Piccolo L, Rimondini M, Rossi A, Carta A, Porru S, Amaddeo F, Lasalvia A. Effectiveness of a Mindful Compassion Care Program in reducing burnout and psychological distress amongst frontline hospital nurses during the COVID-19 pandemic: a study protocol for a randomized controlled trial. Trials. 2022 Sep 2;23(1):734. doi: 10.1186/s13063-022-06666-2. PMID 36056401